CLINICAL TRIAL: NCT01064882
Title: Safety and Efficacy of Bimatoprost Ophthalmic Solution in Increasing Eyelash Prominence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 192024-051
Record Dates: First submitted 2010-02-05; First posted 2010-02-09 (Estimated); Results first posted 2011-12-09 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-11

CONDITIONS: Eyelash Hypotrichosis
MeSH Terms: interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- bimatoprost ophthalmic solution 0.005% (Experimental): bimatoprost ophthalmic sterile solution 0.005%
  Interventions: Drug: bimatoprost ophthalmic solution 0.005%
- bimatoprost ophthalmic solution 0.015% (Experimental): bimatoprost ophthalmic sterile solution 0.015%
  Interventions: Drug: bimatoprost ophthalmic solution 0.015%
- bimatoprost ophthalmic solution 0.03% (Active Comparator): bimatoprost ophthalmic solution 0.03%
  Interventions: Drug: bimatoprost ophthalmic solution 0.03%

INTERVENTIONS:
Drug: bimatoprost ophthalmic solution 0.005% — One drop applied to a sterile single-use-per-eye applicator and applied to upper eyelid margins (where the eyelashes meet the skin)
  Arms: bimatoprost ophthalmic solution 0.005%
Drug: bimatoprost ophthalmic solution 0.015% — One drop applied to a sterile single-use-per-eye applicator and applied to upper eyelid margins (where the eyelashes meet the skin)
  Arms: bimatoprost ophthalmic solution 0.015%
Drug: bimatoprost ophthalmic solution 0.03% — One drop applied to a sterile single-use-per-eye applicator and applied to upper eyelid margins (where the eyelashes meet the skin)
  Other Names: LATISSE®
  Arms: bimatoprost ophthalmic solution 0.03%

SUMMARY:
This study will evaluate the safety and efficacy of bimatoprost ophthalmic solution 0.005% or 0.015% compared with bimatoprost ophthalmic solution 0.03% once-daily application to the upper eyelid margins in increasing eyelash prominence

ELIGIBILITY:
Inclusion Criteria:

* Female Caucasians between 30 and 55 years of age, with hypotrichosis (inadequate or not enough) of the eyelashes
* Eyelash prominence assessment of minimal or moderate

Exclusion Criteria:

* Any eye disease or abnormality
* Any permanent eyeliner or eyelash implants of any kind
* Any ocular surgery, semi-permanent eyelash tint, or eyelash extension application during the 3 months prior to study entry
* Any use of prescription eyelash growth products
* Any use of over the counter eyelash growth products during the 6 months prior to baseline
* Any use of treatments that may affect hair growth during the 6 months prior to baseline

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost Ophthalmic Solution 0.005% | Bimatoprost Ophthalmic Solution 0.015% | Bimatoprost Ophthalmic Solution 0.03%
Started | 36 | 34 | 34
Completed | 34 | 32 | 32
Not Completed | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost Ophthalmic Solution 0.005% | Bimatoprost Ophthalmic Solution 0.015% | Bimatoprost Ophthalmic Solution 0.03% | Total
Number analyzed (Participants) | 36 | 34 | 34 | 104
Age Continuous [Mean (Full Range); unit: years] | 46.9 [32 to 55] | 45.4 [33 to 55] | 46.7 [31 to 55] | 46.3 [31 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 34 | 104
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Eyelash Length at Month 3
Description: Change from Baseline at Month 3 in eyelash length, measured in millimeters (mm). Data from both eyes were averaged for each subject for analysis. Changes from baseline represented by positive values indicated longer length, and changes from baseline represented by negative values indicated shorter length.
Time Frame: Baseline, Month 3
Population: Modified Intent-to-Treat: All randomized (started study) subjects who were treated with the intended study medication and completed at least one-follow-up visit. (Note that one subject in the Bim 0.015% treatment group did not have baseline or Month 3 visit data for this outcome measure.)
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Bimatoprost Ophthalmic Solution 0.005% | Bimatoprost Ophthalmic Solution 0.015% | Bimatoprost Ophthalmic Solution 0.03%
Number analyzed (Participants) | 36 | 33 | 34
millimeters (mm)
  Baseline | 5.65 (0.763) | 5.68 (0.613) | 5.95 (0.744)
  Change from Baseline at Month 3 | 0.74 (0.684) | 0.92 (0.668) | 1.36 (0.944)

2. Secondary Outcome: Change From Baseline in Upper Eyelash Thickness at Month 3
Description: Change from baseline in upper eyelash thickness/fullness at Month 3 was measured within 3 preset areas. Eyelash thickness/fullness was assessed across both eyes as an average of the 3 preset areas measured in millimeters squared (mm^2). Changes from baseline to Month 3 represented by positive values indicated increased eyelash thickness, and changes from baseline represented by negative values indicated thinner eyelash thickness.
Time Frame: Baseline, Month 3
Population: Modified Intent-to-Treat: All randomized (started study) subjects who were treated with the intended study medication and completed at least one follow-up visit. (Note that 2 subjects in the Bim 0.015% treatment group did not have baseline or Month 3 visit data for this outcome measure.)
Measure: Mean (Standard Deviation); unit: Millimeters squared (mm^2)
Arm/Group | Bimatoprost Ophthalmic Solution 0.005% | Bimatoprost Ophthalmic Solution 0.015% | Bimatoprost Ophthalmic Solution 0.03%
Number analyzed (Participants) | 36 | 32 | 34
Millimeters squared (mm^2)
  Baseline | 12.75 (5.502) | 14.67 (7.540) | 13.69 (6.753)
  Change from Baseline at Month 3 | 4.50 (4.760) | 5.64 (5.238) | 8.48 (7.387)

3. Secondary Outcome: Change From Baseline in Upper Eyelash Darkness (in Intensity Units) at Month 3
Description: Change from baseline in upper eyelash darkness at Month 3 was determined by lash intensity within the spline (a narrow area approximately 5 pixels wide that bisects the area of interest). Upper eyelash darkness was measured in both eyes and averaged for analysis. Colors ranged from black=0 to white=255. Lower numbers on this continuum indicated darker colors. Therefore, a change from baseline to Month 3 represented by a negative value indicated increased eyelash darkening.
Time Frame: Baseline, Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Bimatoprost Ophthalmic Solution 0.005% | Bimatoprost Ophthalmic Solution 0.015% | Bimatoprost Ophthalmic Solution 0.03%
Number analyzed (Participants) | 36 | 32 | 34
Units on a Scale
  Baseline | 157.14 (22.814) | 154.41 (21.065) | 162.41 (17.321)
  Change from Baseline at Month 3 | -18.75 (23.276) | -26.55 (22.505) | -29.61 (20.443)

4. Secondary Outcome: Percentage of Subjects With a Clinical Response in Overall Eyelash Prominence on the Global Eyelash Assessment (GEA) at Month 3
Description: Percentage of subjects with a clinical response in overall eyelash prominence at Month 3 was measured using a 4-point GEA scale with the aid of the photonumeric guide. The scale ranges from 1 (minimal = worst) prominence to 4 (very marked = best)prominence. Eyelash prominence was assessed and graded by the investigator over both eyes. A clinical response was defined as at least a 1-grade increase in GEA score from baseline to Month 3.
Time Frame: Month 3
Population: Modified Intent-to-Treat: All randomized (started study) subjects who were treated with the intended study medication and completed at least one follow-up visit.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Bimatoprost Ophthalmic Solution 0.005% | Bimatoprost Ophthalmic Solution 0.015% | Bimatoprost Ophthalmic Solution 0.03%
Number analyzed (Participants) | 36 | 34 | 34
Percentage of Subjects | 52.8 | 79.4 | 85.3

5. Secondary Outcome: Change From Baseline in Overall Eyelash Satisfaction at Month 3
Description: Change from baseline at Month 3 in question 3 "overall, how satisfied are you with your eyelashes?" Responses ranged from 1 (very unsatisfied = worst) to 5 (very satisfied = best). Individual responses at Month 3 were compared to baseline. Positive values at Month 3 indicated an improvement from baseline, and negative values indicated a worsening from baseline.
Time Frame: Baseline, Month 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Bimatoprost Ophthalmic Solution 0.005% | Bimatoprost Ophthalmic Solution 0.015% | Bimatoprost Ophthalmic Solution 0.03%
Number analyzed (Participants) | 36 | 34 | 34
Scores on a Scale
  Baseline | 1.47 (0.560) | 1.56 (0.613) | 1.71 (0.524)
  Change from Baseline at Month 3 | 1.35 (1.323) | 2.25 (1.368) | 2.06 (0.840)

6. Secondary Outcome: Change From Baseline in the Confidence, Attractiveness, and Professionalism (CAP) Domain Scores at Month 3
Description: Change from baseline in the CAP domain at Month 3 included responses to questions 7, 8, and 9. Responses to each question ranged from 1 (very much disagree = worst) to 5 (very much agree = best) with the minimum sum of the scores for the domain equal to 3 and the maximum sum of the scores for the domain equal to 15. Domain responses at Month 3 were compared to baseline. Positive values at Month 3 indicated an improvement from baseline, and negative values indicated a worsening from baseline.
Time Frame: Baseline, Month 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Bimatoprost Ophthalmic Solution 0.005% | Bimatoprost Ophthalmic Solution 0.015% | Bimatoprost Ophthalmic Solution 0.03%
Number analyzed (Participants) | 36 | 34 | 34
Scores on a Scale
  Baseline | 4.33 (2.098) | 4.53 (1.830) | 4.94 (2.029)
  Change from Baseline at Month 3 | 2.79 (3.198) | 4.72 (3.752) | 3.06 (2.526)

7. Secondary Outcome: Treatment Satisfaction Questionnaire Score at Month 3
Description: The Treatment Satisfaction Questionnaire at Month 3 consisted of 2 questions that collected information regarding subject satisfaction with the treatment overall. The questions assessed the likelihood that the subject would use the product, as well as the likelihood that the subject would recommend the product to family and/or friends, if it were available. The score was based on the responses to each question. Questions were answered on a 5-point scale ranging from 1 (very unlikely = worst) to 5 (very likely = best).
Time Frame: Month 3
Population: Modified Intent-to-Treat: All randomized subjects who were treated with the intended study medication and completed at least one follow-up visit.(Note: 2 subjects in the Bim 0.015% treatment group, 1 subject in the Bim 0.005% treatment group, and 1 subject in the Bim 0.03% treatment group did not have Month 3 visit data for this outcome measure)
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Bimatoprost Ophthalmic Solution 0.005% | Bimatoprost Ophthalmic Solution 0.015% | Bimatoprost Ophthalmic Solution 0.03%
Number analyzed (Participants) | 35 | 32 | 33
Scores on a Scale
  If Avail, How Likely Would You Continue to Use It? | 4.1 (1.21) | 4.2 (1.14) | 4.1 (0.93)
  If Avail, How Likely Would You Recommend It? | 4.1 (1.26) | 4.2 (1.07) | 4.4 (0.61)

ADVERSE EVENTS:
Arm/Group | Bimatoprost Ophthalmic Solution 0.005% | Bimatoprost Ophthalmic Solution 0.015% | Bimatoprost Ophthalmic Solution 0.03%
Serious Adverse Events (participants affected / at risk) | 0/36 | 1/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/36 | 7/34 | 2/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost Ophthalmic Solution 0.005% (N=36) | Bimatoprost Ophthalmic Solution 0.015% (N=34) | Bimatoprost Ophthalmic Solution 0.03% (N=34)
Appendicitis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost Ophthalmic Solution 0.005% (N=36) | Bimatoprost Ophthalmic Solution 0.015% (N=34) | Bimatoprost Ophthalmic Solution 0.03% (N=34)
Eyelids Pruritus (Eye disorders) | 0 | 3 | 2
Eyelid Pain (Eye disorders) | 0 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo